CLINICAL TRIAL: NCT03562858
Title: Post-operative Hyper-sensitivity Assessment After Immediate Versus Delayed Dentine Sealing in Teeth for Indirect Tooth Colored Restorations: Randomized Controlled Clinical Trial
Brief Title: Post-operative Hyper-sensitivity Assessment After Immediate Versus Delayed Dentine Sealing in Teeth for Indirect Tooth Colored Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hoda omar tawfeek hussien fouda, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-05-21
Record Dates: First submitted 2018-05-16; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hypersensitivity Dentin
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed dentine sealing (Active Comparator)
  Interventions: Procedure: Delayed dentin sealing protocol
- Immediate dentin sealing (Experimental)
  Interventions: Procedure: Immediate dentin sealing protocol

INTERVENTIONS:
Procedure: Immediate dentin sealing protocol — Sealing of the dentin before impression taking directly after cavity preparation to prevent postoperative hypersensitivity during provisionalization and after cementation
  Arms: Immediate dentin sealing
Procedure: Delayed dentin sealing protocol — Sealing the dentin just prior to cementation
  Arms: Delayed dentine sealing

SUMMARY:
PICOT elements:P: Teeth restored with indirect tooth colored restoration I: Immediate dentin sealing using universal adhesive C: Delayed dentin sealing O: Post-operative Hypersensitivity T: -Hypersensitivity assessment one week during provisionalization period and post-cementation S: Randomized Controlled Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Extensive carious lesions indicated for indirect restorations
* Lower first molars
* Age of patients range is 18 -50 years
* Patients have not received antibiotic therapy for 1 month before sampling
* Males or Females (Both genders)
* Patients with Good oral hygiene
* Co-operative patients approving the trial

Exclusion Criteria:

* Pregnancy
* Systemic disease or severe medical
* Patients having complications as:

Periodontal problems Mobile teeth, arrest caries and non-vital teeth

* Heavy smoking patients
* Xerostomia
* Lack of compliance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative hypersensitivity at baseline | 10 minutes
  The post-operative hypersensitivity assessment will be performed at baseline , using visual analogue scale (VAS) for both intervention and control group . The visual analogue scale is a scale numbered from zero to 10 , where as the range from zero to three resembles from no to very mild sensitivity , the range from four to seven resembles moderate sensitivity and from eight to ten resembles severe sensitivity
Post-operative hypersensitivity one week after temporization | 1 week
  The post-operative hypersensitivity will be assessed one week after temporization for both intervention and control group using the visual analogue scale VAS .The visual analogue scale is a scale numbered from zero to 10 , where as the range from zero to three resembles from no to very mild sensitivity , the range from four to seven resembles moderate sensitivity and from eight to ten resembles severe sensitivity
Post-operative hypersensitivity after cementation of the indirect tooth coloured restoration | 1 week
  The post-operative hypersensitivity will be assessed using visual analogue scale VAS 1 week after cementation of the indirect tooth coloured restoration. The visual analogue scale is a scale numbered from zero to 10 , where as the range from zero to three resembles from no to very mild sensitivity, the range from four to seven resembles moderate sensitivity and from eight to ten resembles severe sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt